CLINICAL TRIAL: NCT03406286
Title: Post-Marketing Surveillance(PMS) of Safety and Efficacy of Samsca® Tablets in Korean Patients With ADPKD
Brief Title: Samsca PMS in ADPKD Patients
Status: Completed | Type: Observational
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 156-402-00110
Record Dates: First submitted 2017-12-22; First posted 2018-01-23 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Safety
Keywords: Post Marketing Surveillance
MeSH Terms: interventions — Tolvaptan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: Tolvaptan
  Other Names: Samsca

SUMMARY:
This is a Post-Marketing Surveillance study(PMS) of Samsca® tablets in actual use in cases to slow the progression of cyst development and renal insufficiency in accordance with Korean regulations on Risk Management Plan(RMP) and New Drug Re-examination. This survey is a post-marketing, prospective, single-arm, all-cases survey conducted on approved indication, usage, dosage.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older patients with CKD(chronic kidney disease) stage 1 to 4 at initiation of treatment with evidence of rapidly progressing disease.
2. Patients who need to be prescribed by Investigators who got registered in Risk Management Plan.
3. Patients who have agreed and signed on conditions specified in Risk Management Plan.

Exclusion Criteria:

1. Patients with known or suspected hypersensitivity to tolvaptan or chemically related structures such as benzazepines or to any ingredient of the drug
2. Patients requiring urgent intervention to raise serum sodium acutely.
3. Inability of the patient to sense or appropriately respond to thirst.
4. Hypovolemic hyponatremia
5. Concomitant use of strong CYP3A(Cytochrome P450, family3, subfamily A) inhibitors
6. Anuric patients
7. Volume depletion patients
8. Hypernatremia patients
9. Women who are pregnant or possibly pregnant and lactation
10. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
11. Patients who are applicable to permanent discontinuation criteria prior to initiation of Samsca® Tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 600 patients will be enrolled for survey period (10 years). Especially, Liver injury cases of all patients in actual use of Samsca® Tablets to slow the progression of cyst development and renal insufficiency will be focused on monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 2067 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
The incidence rate and the number of Adverse Events (AE) / Adverse Drug Response (ADR) | 10 years
  All adverse events (AEs) observed during/after the administration will be analyzed as safety assessment. The number of patients and the number of AE, ADR, Serious AE·ADR, Unexpected AE·ADR will be calculated (frequency and percentage).

CONTACTS AND LOCATIONS:
Locations (1):
- Kim Med Clinic, Ulsan, Gyeongsangnam-do, South Korea